CLINICAL TRIAL: NCT04689360
Title: An Intermediate Size Expanded Access Protocol of Elamipretide for Subcutaneous Injection in Patients With Genetically Confirmed Rare Diseases With Known Mitochondrial Dysfunction
Brief Title: An Intermediate Size Expanded Access Protocol of Elamipretide
Status: Available | Type: Expanded Access
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SPIES-006; SPIES-007 (Other: StealthBiotherapeutics)
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Mitochondrial Diseases; Barth Syndrome
Keywords: Barth
MeSH Terms: conditions — Mitochondrial Diseases; Barth Syndrome | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: elamipretide — Elamipretide is an aromatic-cationic tetrapeptide that readily penetrates cell membranes and transiently localizes to the inner mitochondrial membrane.
  Other Names: MTP-131

SUMMARY:
Choosing to participate in an expanded access program is an important personal decision. Talk with your doctor to learn more about this program. The treating physician must contact StealthBiotherapeutics using the Expanded Access Program Contacts provided. Elamipretide will only be made available after careful review of an individual request submitted by the treating physician. The initiation and conduct of the treatment with elamipretide for an individual patient, and compliance with this treatment guideline, will be under the full and sole responsibility of the treating physician.

ELIGIBILITY:
Key Inclusion Criteria:

1. ≥1 year and ≤ 80 years of age or ≥12 years for Barth Syndrome in SPIES-007
2. Patients with genetically confirmed rare primary mitochondrial diseases including Barth Syndrome

   1. observed cardiomyopathy, renal impairment, neuropathic, or ophthalmic manifestation
   2. where such disease is serious or life-threatening and no comparable or satisfactory alternative therapy options available.
3. Patients without genetic confirmation of a rare disease with known mitochondrial dysfunction but do exhibit serious or life-threatening clinical manifestations of mitochondrial dysfunction.
4. Is self-able or has caregiver willing and able to administer SC injection.
5. Would potentially benefit from treatment with elamipretide and cannot be treated satisfactorily with any approved medicinal product in the opinion of the treating physician.

Key Exclusion Criteria:

1. Known hypersensitivity to elamipretide or any excipients.
2. Women who are pregnant, are planning on becoming pregnant, or are breast-feeding.
3. Patients receiving any other investigational agent within 30 days of dosing.
4. Any active, serious psychiatric, medical, or other conditions/situations which, in the treating physician's opinion, could compromise the patient's safety.

Ages: 1 Year to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult